CLINICAL TRIAL: NCT06286982
Title: Oral Symptoms in Older Patients With Frailty: a Prospective Observational Study Using the Oral Symptom Assessment Scale
Brief Title: The Oral Symptom Assessment Scale in Older Patients With Frailty
Status: Completed | Type: Observational
Sponsor: Our Lady's Hospice and Care Services (Other)
Responsible Party: Principal Investigator, Prof Andrew Davies, Professor, Our Lady's Hospice and Care Services
Other Study IDs: OASIS III
Record Dates: First submitted 2023-08-17; First posted 2024-02-29 (Actual); Last update posted 2025-08-11 (Actual); Status verified 2025-06

CONDITIONS: Frailty; Older Adults
Keywords: Frailty; Mouth; Symptom assessment; Aged
MeSH Terms: conditions — Frailty

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- People aged 65 years and older with a Clinical Frailty Score (CFS) ≥5: The Oral Symptom Assessment Scale will be administered to participants. A feedback questionnaire will also be administered.
  Interventions: Other: Oral Symptom Assessment Scale

INTERVENTIONS:
Other: Oral Symptom Assessment Scale — The Oral Symptom Assessment Scale is a patient-rated oral (or mouth) symptom assessment tool

SUMMARY:
Oral (or mouth) symptoms are common in older patients who live with frailty. It is known that frailty describes someone's overall resilience and how this relates to the chances of recovery following a health problem. A questionnaire called the Oral Symptom Assessment Scale (or OSAS) was designed to look at mouth symptoms in patients who had an advanced cancer. These symptoms may overlap with patients who have frailty.

This research study is taking place to find out if the OSAS will be a suitable questionnaire that can be used in older patients with frailty.

This study will take place in Our Lady's Hospice & Care Services, Harold's Cross and St James' Hospital over six months.

DETAILED DESCRIPTION:
Participants will be asked by one of our researchers about the presence or absence of 21 mouth symptoms in the last week. If present, the participant will be asked about how bothersome each symptom is as well as the severity and frequency. Up to three additional mouth symptoms that are not listed in the OSAS can be reported and rated in the same way by the participant. Participants will be asked about the questionnaire itself to provide feedback. This will take approximately 10-15 minutes to complete both.

ELIGIBILITY:
Inclusion Criteria

* Age ≥ 65 years old
* Clinical Frailty Score ≥ 5
* No known history of dementia
* The attending clinician should have no concerns about a participant's capacity to consent for this research

Exclusion Criteria:

* Inability to provide informed consent
* Inability to complete the questionnaire
* Abbreviated Mental Test Score -4 (AMT4) <4

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: Participants will be patients aged 65 years and older with a Clinical Frailty Score (CFS) ≥5 (as determined by the multi-disciplinary clinical team).
Sampling Method: Non-Probability Sample
Enrollment: 250 (Actual)
Dates: Start 2023-06-06 (Actual); Primary Completion 2025-07-04 (Actual); Study Completion 2025-07-04 (Actual)

PRIMARY OUTCOMES:
To determine the prevalence of oral symptoms in older patients with frailty | In the previous 1 week
  This will be determined by participants indicating the presence ( or absence) of any one of twenty-one oral symptoms on the oral symptom assessment scale.(OSAS).
To determine the clinical features of these oral symptoms in this group (i.e. frequency, severity and level of distress) | In the previous 1 week
  If a participant indicates the presence of an oral symptom, they are asked to rate the frequency (rated : rarely (1), occasionally (2), frequently (3), almost constantly) (4), severity (rated: slight (1), moderate (2), severe (3), very severe (4)) and level of distress (rated: not at all (0.8), a little bit (1.6), somewhat (2.4), quite a bit (3.2), very much (4)) caused by each symptom. The higher the rating, the higher the frequency, severity or distress.
To determine the relationship between oral symptoms and Clinical Frailty Score / Cumulative Illness Rating Scale for Geriatrics/Medications | In the previous 1 week
  The Clinical Frailty Score (CFS) is a clinician-rated single-item written and visual chart with nine graded illustrations. The baseline of the participant in the two weeks prior to presentation should form the basis of the score as opposed to the current, immediate presentation findings. The frailty cut-off point is ≥ 5. It involves the evaluation of domains including cognition, function, and co-morbidity to produce the score. The Cumulative Illness Rating Scale for Geriatrics (CIR-G)is a scale designed to rate both the presence and severity of a disease in older persons. It encompasses information about both the long-term course and as well as current severity of a disease. It is acquired from patient medical records, interviews with patients as well as contemporaneous examination and test findings. A medication list (both regular and as needed medications) will be recorded.
To provide initial validation of OSAS in older patients with frailty | In the previous 1 week
  OSAS refers to the Oral Symptom Assessment Scale - this a twenty item patient-rated oral symptom assessment instrument which was designed and has been validated in patients with advanced cancer. The symptom of 'drooling' will be added based on investigator experience. The rating system has been outlined above.

CONTACTS AND LOCATIONS:
Overall Officials: Davies Andrew, MB MD FRCP, Principal Investigator — Academic Department of Palliative Medicine, Our Lady's Hospice and Care Services, Dublin
Locations (2):
- Ireland (2):
  - St James's Hospital, Dublin, Dublin
  - Our Lady's Hospice and Care Services, Dublin, Dublin

IPD SHARING:
Plan to Share IPD: No
The approved study protocol excludes the sharing of individual participant data with other researchers

REFERENCES:
- [Background] Lindroos EK, Saarela RKT, Suominen MH, Muurinen S, Soini H, Kautiainen H, Pitkala KH. Burden of Oral Symptoms and Its Associations With Nutrition, Well-Being, and Survival Among Nursing Home Residents. J Am Med Dir Assoc. 2019 May;20(5):537-543. doi: 10.1016/j.jamda.2018.10.025. Epub 2018 Dec 9. PMID 30541688
- [Background] Saarela RKT, Savikko NM, Soini H, Muurinen S, Suominen MH, Kautiainen H, Pitkala KH. Burden of Oral Symptoms and Health-Related Quality of Life in Long-Term Care Settings in Helsinki, Finland. J Nutr Health Aging. 2019;23(10):1021-1025. doi: 10.1007/s12603-019-1268-9. PMID 31781733
- [Background] Miller MD, Paradis CF, Houck PR, Mazumdar S, Stack JA, Rifai AH, Mulsant B, Reynolds CF 3rd. Rating chronic medical illness burden in geropsychiatric practice and research: application of the Cumulative Illness Rating Scale. Psychiatry Res. 1992 Mar;41(3):237-48. doi: 10.1016/0165-1781(92)90005-n. PMID 1594710
- [Background] Locke T, Keat S, Tate M, Bown A, Hart A, Ghosh R. Assessing the performance of the four question abbreviated mental test in the acute geriatric setting. Acute Med. 2013;12(1):13-7. PMID 23539371
- [Background] Davies A, Buchanan A, Todd J, Gregory A, Batsari KM. Oral symptoms in patients with advanced cancer: an observational study using a novel oral symptom assessment scale. Support Care Cancer. 2021 Aug;29(8):4357-4364. doi: 10.1007/s00520-020-05903-1. Epub 2021 Jan 8. PMID 33416995
- [Background] Fried LP, Ferrucci L, Darer J, Williamson JD, Anderson G. Untangling the concepts of disability, frailty, and comorbidity: implications for improved targeting and care. J Gerontol A Biol Sci Med Sci. 2004 Mar;59(3):255-63. doi: 10.1093/gerona/59.3.m255. PMID 15031310